CLINICAL TRIAL: NCT03322566
Title: A Randomized Phase 2 Study of the Combination of Pembrolizumab (MK-3475) Plus Epacadostat (INCB024360) With Platinum-based Chemotherapy Versus Pembrolizumab Plus Platinum-based Chemotherapy Plus Placebo as First-Line Treatment in Patients With Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study of Pembrolizumab Plus Epacadostat With Platinum-based Chemotherapy Versus Pembrolizumab Plus Platinum-based Chemotherapy Plus Placebo in Metastatic Non-Small Cell Lung Cancer (KEYNOTE-715-06/ECHO-306-06)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KEYNOTE-715-06/ECHO-306-06; 2017-001810-27 (EudraCT Number)
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Results first posted 2020-01-29 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Lung Cancer
Keywords: Non-small cell lung cancer; programmed cell death 1 (PD-1) inhibitor; indoleamine 2; 3-dioxygenase 1 (IDO1) inhibitor; chemotherapy
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; epacadostat; Platinum Compounds

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pembrolizumab + Chemotherapy + Epacadostat (Experimental): Participant received pembrolizumab 200 mg intravenous (IV) infusion, every 3 weeks (Q3W) on Day 1 of each 21 day cycle for up to 35 cycles + epacadostat 100 mg tablets, orally, twice daily (BID) in each 21 day cycle for up to 35 cycles + platinum-doublet chemotherapy (pemetrexed 500 mg/m^2 IV infusion, Q3W + cisplatin 75 mg/m^2 IV infusion, Q3W or carboplatin 5-6 mg/mL/min IV infusion Q3W for 4 cycles followed by pemetrexed maintenance; or paclitaxel 200 mg /m^2 IV infusion, Q3W + carboplatin 5-6 mg/mL/min IV infusion Q3W for 4 cycles).
  Interventions: Drug: Pembrolizumab; Drug: Epacadostat; Drug: Platinum-based chemotherapy
- Pembrolizumab + Chemotherapy + Placebo (Experimental): Participant received pembrolizumab 200 mg IV infusion, Q3W on Day 1 of each 21 day cycle for up to 35 cycles + epacadostat matching placebo tablets, orally, BID in each 21 day cycle for up to 35 cycles + platinum-doublet chemotherapy (pemetrexed 500 mg/m^2 IV infusion, Q3W + cisplatin 75 mg/m^2 IV infusion, Q3W or carboplatin 5-6 mg/mL/min IV infusion Q3W for 4 cycles followed by pemetrexed maintenance; or paclitaxel 200 mg /m^2 IV infusion, Q3W + carboplatin 5-6 mg/mL/min IV infusion Q3W for 4 cycles).
  Interventions: Drug: Pembrolizumab; Drug: Platinum-based chemotherapy; Drug: Placebo
- Pembrolizumab + Epacadostat (Experimental): Participant received pembrolizumab 200 mg IV infusion, Q3W on Day 1 of each 21 day cycle for up to 35 cycles + epacadostat 100 mg tablets, orally, BID in each 21 day cycle for up to 35 cycles.
  Interventions: Drug: Pembrolizumab; Drug: Epacadostat

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab administered intravenously every 3 weeks.
  Other Names: MK-3475
Drug: Epacadostat — Epacadostat administered orally twice daily.
  Other Names: INCB024360
  Arms: Pembrolizumab + Chemotherapy + Epacadostat; Pembrolizumab + Epacadostat
Drug: Platinum-based chemotherapy — Investigator selected one of the following regimens: pemetrexed + cisplatin, pemetrexed + carboplatin, or paclitaxel + carboplatin, depending on histology.
  Arms: Pembrolizumab + Chemotherapy + Epacadostat; Pembrolizumab + Chemotherapy + Placebo
Drug: Placebo — Matching placebo administered orally twice daily.
  Arms: Pembrolizumab + Chemotherapy + Placebo

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of pembrolizumab plus epacadostat with platinum-based chemotherapy versus pembrolizumab plus platinum-based chemotherapy plus placebo as first-line therapy in participants with metastatic non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of stage IV NSCLC without epidermal growth factor receptor (EGFR)-sensitizing mutation, ROS1 and/or anaplastic lymphoma kinase (ALK) translocation
* Measurable disease based on RECIST 1.1
* Life expectancy of at least 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function per protocol-defined criteria.
* Provide tumor tissue sample.

Exclusion Criteria:

* Known untreated central nervous system metastases and/or carcinomatous meningitis
* History of (non-infectious) pneumonitis that required systemic steroids or current pneumonitis/interstitial lung disease.
* Symptomatic ascites or pleural effusion.
* Known history of an additional malignancy, except if the participant has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy.
* Active autoimmune disease that has required systemic treatment in past 2 years.
* Has had an allogeneic tissue/solid organ transplant.
* Has a known history of human immunodeficiency virus (HIV) infection. HIV testing is not required unless mandated by the local health authority.
* Has known history of or is positive for active Hepatitis B (HBsAg reactive) or has active Hepatitis C (HCV RNA). Note: Testing must be performed to determine eligibility.
* History or presence of an abnormal electrocardiogram (ECG) that, in the Investigator's opinion, is clinically meaningful.
* Use of protocol-defined prior/concomitant therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2020-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lance Leopold, MD, Study Director — Incyte Corporation
Locations (94):
- United States (21):
  - Southern Cancer Center, PC, Daphne, Alabama
  - Western Regional Medical Center, Inc., Goodyear, Arizona
  - Arizona Oncology Associates PC- HOPE, Tucson, Arizona
  - Lynn Cancer Institute, Boca Raton, Florida
  - Florida Cancer Specialists (South Region), Fort Myers, Florida
  - Florida Cancer Specialists (North Region), St. Petersburg, Florida
  - PPG-Oncology, Fort Wayne, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - MMCORC, Saint Louis Park, Minnesota
  - St. Vincent Healthcare Frontier Cancer Center, Billings, Montana
  - New York Oncology Hematology P.C, Albany, New York
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Southwestern Regional Medical Center, Inc., Tulsa, Oklahoma
  - St. Luke's Hospital - Anderson Campus, Easton, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Tennessee Oncology, PLLC/The Sarah Cannon Research Institute, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC/The Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology-Denton South, Denton, Texas
  - Oncology & Hematology Assoc. SW Virginia, Inc., DBA Blue Ridge Cancer Care, Blacksburg, Virginia
  - Emily Couric Clinical Cancer Center, Charlottesville, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (6):
  - Blacktown Hospital, Blacktown, New South Wales
  - Chris OBrien Lifehouse, Camperdown, New South Wales
  - The Crown Princess Mary Cancer Centre Westmead, Westmead, New South Wales
  - Southern Medical Day Care Centre, Wollongong, New South Wales
  - MNCCI Port Macquarie Base Hospital, Port Macquarie, New South Wales (Australia)
  - Cairns Base Hospital, Cairns, Queensland
- Canada (8):
  - BCCA-Cancer Centre of the Southern Interior, Kelowna, British Columbia
  - Lions Gate Hospital, North Vancouver, British Columbia
  - CISSS de la Monteregie-Centre, Greenfield Park, Quebec
  - CSSS de Laval- Hopital de la Cite de la Sante, Laval, Quebec
  - CIUSSS Ouest de l'Ile - St-Mary's Hospital, Montreal, Quebec
  - CIUSSS du Nord-de-l'ILe-de-Montreal Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - CHU de Quebec - Hotel-Dieu de Quebec, Québec, Quebec
  - CIUSSS de la Mauricie-et-du-Centre-du-Quebec, Trois-Rivières, Quebec
- Hungary (6):
  - Zala Megyei Korhaz Pozvai Telephely, Pózva, Zalaegerszeg
  - Orszagos Koranyi TBC es Pulmonologiai Intezet, Budapest
  - Veszprem Megyei Tudogyogyintezet, Farkasgyepű
  - Bekes Megyei Pandy Kalman Korhaz, Gyula
  - CRU Hungary Kft., Miskolc
  - Jasz Nagykun Szolnok Megyei Hetenyi Geza Korhaz Rendelointezet, Szolnok
- St Vincents University Hospital, Dublin, Ireland
- Israel (6):
  - Ha Emek Medical Center, Afula
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medcal Center, Ramat Gan
- Italy (5):
  - Centro Di Riferimento Oncologico, Aviano
  - A.O.U. Policlinico Vittorio Emanuele - Presidio Gaspare Rodolico, Catania
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Europeo di Oncologia, Milan
  - Ospedale San Gerardo - ASST Monza, Monza
- Mexico (3):
  - Medical Care Research S.A. de C.V., Mérida, Yucatán
  - Oaxaca Site Management Organization S.C., Oaxaca City
  - FAICIC Clinical Research, Veracruz
- Russia (10):
  - Belgorod Regional Oncology Dispensary, Belgorod
  - Udmurtia Republic Regional Clinical Oncology Dispensary, Izhevsk
  - Republican Clinical Oncology Dispensary of Tatarstan MoH, Kazan'
  - Central Clinical Hospital with polyclinic, Moscow
  - Moscow Research Oncology Institute, Moscow
  - SBI of Stavropol region Pyatigorskiy Oncologic dispensary, Pyatigorsk
  - SBHI Leningrad Regional Clinical Hospital, Saint Petersburg
  - SBHI Samara Regional Clinical Oncology Dispensary, Samara
  - Oncological Dispensary #2 of Ministry of Health of Krasnodar region, Sochi
  - Tomsk Scientific Research Institute of Oncology, Tomsk
- South Korea (4):
  - National Cancer Center, Goyang-si
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria, Gran Canaria
  - Hospital Juan Ramón Jimenez, Huelva
  - Institut Catala Oncologia de Bellvitge - ICO, L'Hospitalet de Llobregat
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario La Fe, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- Taiwan (5):
  - Chang Gung Medical Foundation, Kaohsiung Branch, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation, Linkou Branch, Taoyuan District
- Turkey (Türkiye) (9):
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir, Bornova
  - Baskent Universitesi Adana Uygulama ve Arastirma Hastanesi, Adana
  - Cukurova Universitesi Tıp Fakultesi Balcalı Hastanesi, Adana
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Uludag Universitesi Tip Fakultesi, Bursa
  - Pamukkale Unv. Tip Fak, Denizli
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Samsun Medical Park Hastanesi, Samsun
  - Namık Kemal University Medical Faculty, Tekirdağ
- United Kingdom (4):
  - Mount Vernon Cancer Centre, Northwood, Middlesex
  - Western General Hospital, Edinburgh
  - North Middlesex Hospital, London
  - Freeman Hospital Newcastle upon Tyne Foundation NHS Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boyer M, Hui R, Urban D, Clingan P, Su WC, Devaux C, Gadgeel S, Garassino M, Leopold L, Daniel J, Munteanu MC, Samkari A, Luo Y, Abreu DR. Pembrolizumab with platinum-based chemotherapy with or without epacadostat as first-line treatment for metastatic non-small cell lung cancer: a randomized, partially double-blind, placebo-controlled phase II study. BMC Cancer. 2024 Jul 25;23(Suppl 1):1250. doi: 10.1186/s12885-022-10427-4. PMID 39054462

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 65 investigative sites in 14 countries from 09 January 2018 to 13 December 2018.
Pre-assignment Details: Phase 3 design of the study has been amended soon after it had started to a prospectively randomized phase 2 study. At the time of amendment existing participants were given a choice to move/participate in the new phase 2 study, and some participants who chose to discontinue the study at phase 3 were assigned to "study terminated by sponsor" as the reason for not completing the study in disposition table. The results posted are combined in the prospectively redesigned phase 2 trial.
Period: Overall Study
Arm/Group | Pembrolizumab + Chemotherapy + Epacadostat | Pembrolizumab + Chemotherapy + Placebo | Pembrolizumab + Epacadostat
Started | 91 | 87 | 55
Completed | 46 | 42 | 22
Not Completed | 45 | 45 | 33
Not completed — Death | 34 | 35 | 23
Not completed — Physician Decision | 6 | 7 | 2
Not completed — Withdrawal by Subject | 4 | 3 | 6
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Study terminated by sponsor | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were randomized to study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Chemotherapy + Epacadostat | Pembrolizumab + Chemotherapy + Placebo | Pembrolizumab + Epacadostat | Total
Number analyzed (Participants) | 91 | 87 | 55 | 233
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (11.7) | 63.6 (8.8) | 62.8 (8.4) | 63.2 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 30 | 16 | 79
  Male | 58 | 57 | 39 | 154
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian Or Alaska Native | 1 | 0 | 0 | 1
  Race: Asian | 11 | 10 | 2 | 23
  Race: Black Or African American | 1 | 1 | 0 | 2
  Race: White | 78 | 75 | 53 | 206
  Race: Missing | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 3 | 1 | 1 | 5
  Ethnicity: Not Hispanic or Latino | 86 | 85 | 52 | 223
  Ethnicity: Unknown | 2 | 1 | 1 | 4
  Ethnicity: Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) of Pembrolizumab + Chemotherapy + Epacadostat Versus Pembrolizumab + Chemotherapy + Placebo
Description: ORR is defined as the percentage of participants who have a confirmed complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) based on blinded independent central review (BICR).
Time Frame: Assessed every 12 weeks up to 24 months
Population: ITT population consisted of all participants randomized in treatment arm Pembrolizumab+Epacadostat+Chemotherapy and treatment arm Pembrolizumab+Chemothrapy. This is not a primary outcome measure for treatment arm Pembrolizumab+Epacadostat per protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab + Chemotherapy + Epacadostat | Pembrolizumab + Chemotherapy + Placebo
Number analyzed (Participants) | 91 | 87
percentage of participants | 26.4 [17.7 to 36.7] | 44.8 [34.1 to 55.9]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy + Epacadostat vs Pembrolizumab + Chemotherapy + Placebo; Test type: Superiority; p = 0.9948, Stratified Miettinen and Nurminen method — One-sided p-value for testing. H0: difference in % = 0 versus H1: difference in % > 0; Difference in Percentages = -18.5, 95% CI 2-sided [-32.0 to -4.3] — Stratified by PD-L1 TPS ( <50% vs. >=50% ) and predominant tumor histology (squamous vs non-squamous);because of small sample size, the strata 'TPS >= 50 percent Non-squamous' and 'TPS >= 50% Squamous' were combined into one stratum

2. Secondary Outcome: Progression-free Survival of Pembrolizumab + Chemotherapy + Epacadostat Versus Pembrolizumab + Chemotherapy + Placebo
Description: Defined as the time from randomization to the first documented progressive disease (PD) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or death due to any cause, whichever occurs first.
Time Frame: Up to 24 months
Population: ITT population consisted of all participants randomized in treatment arm Pembrolizumab+Epacadostat+Chemotherapy and treatment arm Pembrolizumab+Chemothrapy. This is not a secondary outcome measure for treatment arm Pembrolizumab+Epacadostat per protocol.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab + Chemotherapy + Epacadostat | Pembrolizumab + Chemotherapy + Placebo
Number analyzed (Participants) | 91 | 87
months | 8.0 [4.2 to 10.2] | 8.2 [6.0 to NA] — Upper bound is not estimable
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy + Epacadostat vs Pembrolizumab + Chemotherapy + Placebo; Test type: Other; p = 0.94305, Regression, Cox — One-sided p-value based on log-rank test stratified by TPS (<50% vs >=50%) and predominant histology (squamous vs non-squamous), because of small sample size, the strata 'TPS >= 50% Non-squamous' and 'TPS >= 50% Squamous' were combined into one; Efron's method of tie handling; Hazard Ratio (HR) = 1.47, 95% CI 2-sided [0.91 to 2.36]

3. Secondary Outcome: Overall Survival of Pembrolizumab + Chemotherapy + Epacadostat Versus Pembrolizumab + Chemotherapy + Placebo
Description: Defined as the time from randomization to death due to any cause.
Time Frame: Up to 24 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab + Chemotherapy + Epacadostat | Pembrolizumab + Chemotherapy + Placebo
Number analyzed (Participants) | 91 | 87
months | NA [NA to NA] — Median could not be estimated because there were not enough events | NA [NA to NA] — Median could not be estimated because there were not enough events
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy + Epacadostat vs Pembrolizumab + Chemotherapy + Placebo; Test type: Other; p = 0.96272, Regression, Cox — One-sided p-value based on log-rank test stratified by PD-L1 TPS (<50% vs >=50%) and predominant tumor histology (squamous vs non-squamous), because of small sample size, the strata (<50% vs >=50%) were combined into one stratum; Hazard Ratio (HR) = 1.90, 95% CI 2-sided [0.93 to 3.90]

4. Secondary Outcome: Duration of Response of Pembrolizumab + Chemotherapy + Epacadostat Versus Pembrolizumab + Chemotherapy + Placebo
Description: Defined as the time from the earliest date of qualifying response until earliest date of disease progression, per RECIST v1.1, or death from any cause, whichever comes first.
Time Frame: Up to 24 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab + Chemotherapy + Epacadostat | Pembrolizumab + Chemotherapy + Placebo
Number analyzed (Participants) | 91 | 87
months | NA [1.1 to 7.0] — Median could not be estimated because there were not enough events | 7.0 [1.2 to 8.0]

5. Secondary Outcome: Safety and Tolerability of Pembrolizumab + Chemotherapy + Epacadostat Versus Pembrolizumab + Chemotherapy + Placebo as Measured by the Number of Participants Experiencing Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: Up to 25 months
Population: All Subjects as Treated consists of all randomized participants who received at least one dose of study treatment. This is not a secondary outcome measure for treatment arm Pembrolizumab+Epacadostat per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Chemotherapy + Epacadostat | Pembrolizumab + Chemotherapy + Placebo
Number analyzed (Participants) | 90 | 86
Participants | 89 | 82

6. Secondary Outcome: Safety and Tolerability of Pembrolizumab + Chemotherapy + Epacadostat Versus Pembrolizumab + Chemotherapy + Placebo as Measured by the Number of Participants Discontinuing Study Drug Due to AEs
Description: An AE is defined as any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of any study drug, whether or not considered related to the study drug.
Time Frame: Up to 25 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Chemotherapy + Epacadostat | Pembrolizumab + Chemotherapy + Placebo
Number analyzed (Participants) | 90 | 86
Participants | 37 | 35

ADVERSE EVENTS:
Time Frame: Up to 25 months
Description: All participants as treated (APaT) population included all randomized participants who received at least one dose of study treatment.
Groups:
- Total: Total
Arm/Group | Pembrolizumab + Chemotherapy + Epacadostat | Pembrolizumab + Chemotherapy + Placebo | Pembrolizumab + Epacadostat | Total
All-Cause Mortality (participants affected / at risk) | 38/90 | 35/86 | 26/52 | 99/228
Serious Adverse Events (participants affected / at risk) | 47/90 | 41/86 | 20/52 | 108/228
Other Adverse Events (participants affected / at risk) | 87/90 | 81/86 | 51/52 | 219/228
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Chemotherapy + Epacadostat (N=90) | Pembrolizumab + Chemotherapy + Placebo (N=86) | Pembrolizumab + Epacadostat (N=52) | Total (N=228)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Breakthrough pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 4 (4)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 1 (3)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 2 (2) | 0 (0) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0) | 0 (0) | 5 (5)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gallbladder rupture (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypopharyngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 3 (4) | 1 (1) | 0 (0) | 4 (5)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2) | 8 (8) | 15 (15)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0) | 2 (3)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pancreatic enzymes increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 5 (5)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 12 (12) | 4 (4) | 21 (21)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 4 (4)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Radiation necrosis (Injury, poisoning and procedural complications) | 1 (3) | 1 (1) | 0 (0) | 2 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 4 (4)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Chemotherapy + Epacadostat (N=90) | Pembrolizumab + Chemotherapy + Placebo (N=86) | Pembrolizumab + Epacadostat (N=52) | Total (N=228)
Abdominal pain (Gastrointestinal disorders) | 6 (8) | 3 (3) | 5 (5) | 14 (16)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 7 (8) | 0 (0) | 10 (11)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 6 (6) | 0 (0) | 10 (10)
Alanine aminotransferase increased (Investigations) | 15 (20) | 10 (12) | 1 (3) | 26 (35)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (11) | 16 (16) | 0 (0) | 27 (27)
Amylase increased (Investigations) | 10 (14) | 10 (10) | 7 (8) | 27 (32)
Anaemia (Blood and lymphatic system disorders) | 24 (34) | 37 (56) | 8 (11) | 69 (101)
Anxiety (Psychiatric disorders) | 3 (3) | 5 (5) | 2 (2) | 10 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (21) | 10 (13) | 5 (5) | 29 (39)
Aspartate aminotransferase increased (Investigations) | 15 (22) | 8 (10) | 3 (5) | 26 (37)
Asthenia (General disorders) | 12 (14) | 18 (24) | 6 (9) | 36 (47)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (18) | 10 (10) | 8 (9) | 32 (37)
Blood alkaline phosphatase increased (Investigations) | 7 (7) | 3 (4) | 2 (2) | 12 (13)
Blood creatinine increased (Investigations) | 7 (8) | 7 (11) | 4 (4) | 18 (23)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (8) | 0 (0) | 3 (3) | 8 (11)
Chest pain (General disorders) | 3 (3) | 13 (13) | 10 (11) | 26 (27)
Constipation (Gastrointestinal disorders) | 26 (40) | 23 (35) | 8 (9) | 57 (84)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 11 (13) | 12 (14) | 33 (37)
Decreased appetite (Metabolism and nutrition disorders) | 19 (23) | 20 (23) | 8 (11) | 47 (57)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 2 (2) | 3 (6) | 9 (13)
Diarrhoea (Gastrointestinal disorders) | 23 (36) | 23 (35) | 14 (19) | 60 (90)
Dizziness (Nervous system disorders) | 16 (17) | 13 (17) | 5 (7) | 34 (41)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 5 (5) | 0 (0) | 6 (6)
Dysgeusia (Nervous system disorders) | 8 (9) | 5 (6) | 0 (0) | 13 (15)
Dyspepsia (Gastrointestinal disorders) | 6 (11) | 1 (2) | 3 (5) | 10 (18)
Dysphagia (Gastrointestinal disorders) | 5 (5) | 4 (4) | 0 (0) | 9 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 11 (11) | 7 (7) | 30 (32)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (8) | 1 (1) | 14 (16)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 5 (6) | 1 (1) | 9 (10)
Fatigue (General disorders) | 28 (40) | 25 (32) | 14 (16) | 67 (88)
Gamma-glutamyltransferase increased (Investigations) | 5 (5) | 7 (12) | 3 (3) | 15 (20)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (9) | 3 (3) | 14 (16)
Headache (Nervous system disorders) | 14 (18) | 11 (13) | 5 (7) | 30 (38)
Hypercalcaemia (Metabolism and nutrition disorders) | 5 (6) | 1 (1) | 1 (1) | 7 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (6) | 6 (6) | 2 (5) | 12 (17)
Hypertension (Vascular disorders) | 5 (7) | 3 (4) | 0 (0) | 8 (11)
Hyperthyroidism (Endocrine disorders) | 6 (8) | 6 (6) | 3 (3) | 15 (17)
Hypoaesthesia (Nervous system disorders) | 7 (7) | 7 (8) | 0 (0) | 14 (15)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (3) | 5 (6) | 0 (0) | 6 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (13) | 8 (12) | 1 (1) | 18 (26)
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 (12) | 7 (10) | 1 (1) | 16 (23)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 6 (11) | 1 (1) | 11 (16)
Hypothyroidism (Endocrine disorders) | 10 (10) | 9 (9) | 7 (8) | 26 (27)
Insomnia (Psychiatric disorders) | 16 (16) | 7 (7) | 2 (2) | 25 (25)
Lacrimation increased (Eye disorders) | 11 (13) | 8 (8) | 0 (0) | 19 (21)
Leukopenia (Blood and lymphatic system disorders) | 6 (25) | 4 (7) | 0 (0) | 10 (32)
Lipase increased (Investigations) | 7 (9) | 6 (7) | 5 (5) | 18 (21)
Mucosal inflammation (General disorders) | 5 (7) | 7 (8) | 0 (0) | 12 (15)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3) | 2 (3) | 11 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 2 (2) | 10 (10)
Nasopharyngitis (Infections and infestations) | 5 (8) | 5 (9) | 3 (3) | 13 (20)
Nausea (Gastrointestinal disorders) | 38 (80) | 37 (101) | 10 (13) | 85 (194)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 1 (1) | 8 (8)
Neuropathy peripheral (Nervous system disorders) | 14 (14) | 10 (10) | 1 (2) | 25 (26)
Neutropenia (Blood and lymphatic system disorders) | 16 (24) | 15 (25) | 2 (3) | 33 (52)
Neutrophil count decreased (Investigations) | 4 (8) | 14 (20) | 0 (0) | 18 (28)
Oedema peripheral (General disorders) | 14 (20) | 10 (11) | 4 (4) | 28 (35)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 1 (1) | 8 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (12) | 5 (5) | 2 (3) | 18 (20)
Paraesthesia (Nervous system disorders) | 6 (6) | 1 (1) | 0 (0) | 7 (7)
Peripheral swelling (General disorders) | 6 (9) | 2 (3) | 1 (1) | 9 (13)
Platelet count decreased (Investigations) | 5 (9) | 9 (12) | 0 (0) | 14 (21)
Pneumonia (Infections and infestations) | 7 (7) | 1 (1) | 2 (2) | 10 (10)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (7) | 0 (0) | 8 (9)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 4 (4) | 10 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (13) | 11 (14) | 6 (11) | 29 (38)
Pyrexia (General disorders) | 15 (21) | 10 (12) | 9 (13) | 34 (46)
Rash (Skin and subcutaneous tissue disorders) | 22 (35) | 18 (25) | 10 (13) | 50 (73)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 0 (0) | 7 (7)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 0 (0) | 2 (2) | 12 (14)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (14) | 2 (3) | 0 (0) | 11 (17)
Upper respiratory tract infection (Infections and infestations) | 11 (14) | 6 (7) | 1 (1) | 18 (22)
Urinary tract infection (Infections and infestations) | 5 (8) | 9 (10) | 4 (4) | 18 (22)
Viral infection (Infections and infestations) | 5 (6) | 2 (3) | 0 (0) | 7 (9)
Vomiting (Gastrointestinal disorders) | 19 (29) | 11 (14) | 6 (6) | 36 (49)
Weight decreased (Investigations) | 10 (10) | 8 (9) | 7 (7) | 25 (26)

LIMITATIONS AND CAVEATS:
Data from the final analysis of KEYNOTE-715/ECHO-306 (data cutoff: 13-DEC-2018) indicated that the study did not meet the pre-specified endpoint of improvement in objective response rate (ORR).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT03322566/Prot_SAP_000.pdf